CLINICAL TRIAL: NCT04016038
Title: Sedation in Palliative Care Management Context for Cancer Patients
Brief Title: Psychosocial Approach and Sedation Practices
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-64
Record Dates: First submitted 2019-04-16; First posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: End Stage Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- QualiPas Observational: Prospective qualitative study through a participant observation procedure with 8 care teams practicing within Palliative Care Units, Palliative Care Mobile Team or Territorial Palliative Care Team.
  Interventions: Other: a psycho-social investigation
- QualiPas clinical interview: Qualitative study retrospective research interviews with the doctor and another carer involved in the care of the patient, and close relatives of patients who had sedated before their death. The interviews will be based on 50 cases of patients who have been sedated.
  Interventions: Other: a psycho-social investigation
- QualiPas Focus: Qualitative study by group focus group interviews with clinical teams participating in the project.
  Interventions: Other: a psycho-social investigation

INTERVENTIONS:
Other: a psycho-social investigation — The design of this project is based partly on the UNBIASED international study and is based on an in-depth case study in a prospective and retrospective dimension of deceased cancer patients for whom sedation has been established, and this, during a given period in different care settings: home, care center, hospital and palliative care unit.

SUMMARY:
This study aims to explore deeply the representations and emotional impact of MS on caregivers (doctors and nurses) and relatives of cancer patients. It also aims to describe their collaboration modalities, roles and responsibilities during the decision-making process, implementation and "control" of MS. The project is a multi-center psychosocial study (home, hospitals and palliative care unit) that will take the form of a comprehensive qualitative study, both prospective (participant observation) and retrospective (interview), of patients with and without cancer, for which MS has been administered.

DETAILED DESCRIPTION:
Scientific Background: Physicians have an ethical obligation to relieve the refractory symptoms of patients with advanced cancer. In some situations, in the face of physical symptoms and psycho-existential distress, usual treatment is not effective and palliative sedation (PS) is one of the only acceptable options. The carers, but also the relatives of the patient, are particularly involved in the process of decision-making, information and management of sedation. Despite the interest of MS practice and its impact on different levels (relational, emotional, professional, ethical), and contrary to the important development of international studies in this field, there is a lack of research in France.

Objectives of the project and a brief description of the methods: This study aims to explore in depth the representations and emotional impact of MS on carers (doctors and nurses) and relatives of cancer patients. It also aims to describe their collaboration modalities, roles and responsibilities during the decision-making process, implementation and "control" of MS. The project is a multi-center psychosocial study (home, hospitals and palliative care unit) that will take the form of a comprehensive qualitative study, both prospective (participant observation) and retrospective (interview), of patients with and without cancer, for which MS has been administered.

Expected Outcomes: The expected results are the production of original knowledge about the practice of MS in different clinical settings (hospital, home), a better understanding of the psychosocial determinants of palliative sedation decision-making, an update of knowledge transferable to develop palliative care programs that integrate the experiential, emotional, and contextual dimensions of palliative sedation, a better understanding of the communication skills needed to cope with this practice, and an awareness of health care teams and advocates. public health on this subject.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Anyone from the team during the observation period
* Having accepted the presence of the observer
* Aged over 18

Exclusion Criteria:

* Members of the health care team not present during the observation period
* Member of the team refusing the presence of the observer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the framework of the QualiPaS_OBS study, the observations will be made by a psychologist integrated into each care team during the observations observation period - no professional activity other than observations. The population studied in the QualiPaS_OBS phase corresponds to the members of the health care team practicing within the eight teams of the services participating in the study, as well as secondarily the patients and relatives of the patients concerned by the activity of the team in question. during the observation period.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessing the quality of life | 36 months
  Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Garrido, Study Director — Assistance Publique Hopitaux De Marseille
Locations (2):
- France (2):
  - Assistance des Hôpitaux de Marseille, Marseille
  - Assistance Publique Hopitaux de Marseille, Marseille

REFERENCES:
- [Derived] Vieille M, Dany L, Coz PL, Avon S, Keraval C, Salas S, Bernard C. Perception, Beliefs, and Attitudes Regarding Sedation Practices among Palliative Care Nurses and Physicians: A Qualitative Study. Palliat Med Rep. 2021 May 24;2(1):160-167. doi: 10.1089/pmr.2021.0022. eCollection 2021. PMID 34223516